CLINICAL TRIAL: NCT05274204
Title: Expanded Access to CA102N in One Patient Who Completed at Least 12 Cycles of Combination Therapy of CA102N Plus Lonsurf in Clinical Study Number of HS-CA102N-101
Brief Title: Individual Patient Expanded Access to CA102N
Status: Temporarily not available | Type: Expanded Access
Sponsor: Holy Stone Healthcare Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: HS-CA102N-102
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Advanced or Metastatic Colorectal Cancer (mCRC)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: CA102N
  Other Names: Nim-HA Conjugate

SUMMARY:
This study is an individual patient expanded access protocol that the subject enrolled had completed the combination treatment of CA102N plus Lonsurf for at least 12 cycles.

DETAILED DESCRIPTION:
In the individual patient expanded access, the subject who was enrolled in Phase 1 trial (Study Number: HS-CA102N-101) Part 2 (dose expansion) and had completed at least 12 treatment cycles with CA102N combined with trifluridine /tipiracil (LONSURF) will be provided access to treatment with CA102N (0.72 mg/kg Nimesulide Equivalent of CA102N).

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult